CLINICAL TRIAL: NCT07298512
Title: Clinico-radiological Correlation of MRI Findings in Patients With Temporomandibular Joint Disc Perforation
Acronym: TMJ Disc
Status: Completed | Type: Observational
Sponsor: Recep Tayyip Erdogan University Training and Research Hospital (Other)
Responsible Party: Principal Investigator, DİLARA NİL GÜNAÇAR, Assoc. Prof., Recep Tayyip Erdogan University Training and Research Hospital
Other Study IDs: 2025/48
Record Dates: First submitted 2025-12-03; First posted 2025-12-23 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Temporomandibular Joint Disc Displacement; Magnetic Resonance Imaging; Bone Marrow

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1: Disc Perforation Group: Participants who demonstrate temporomandibular joint (TMJ) disc perforation on MRI. This cohort will be used to evaluate imaging characteristics and clinical parameters associated with perforation.
- Group 2: Non-Perforation Group: Participants without MRI evidence of TMJ disc perforation.

SUMMARY:
To evaluate the presence of TMJ disc perforation on MRI and investigate its associations with internal disc derangements, disc configuration, condylar bone marrow signal patterns, joint effusion, and demographic or clinical variables such as age, sex, dental status, and pain severity.

DETAILED DESCRIPTION:
This study will prospectively evaluate temporomandibular joint (TMJ) disc perforation using magnetic resonance imaging (MRI) in a diverse adult population. The investigation will focus on identifying the prevalence of disc perforation and examining its relationship with key TMJ structural and functional parameters. Specifically, the study will assess internal disc derangements, variations in disc morphology, condylar bone marrow signal characteristics, and the presence of joint effusion. In addition, demographic and clinical factors-including age, sex, dental status, and pain severity-will be analyzed to determine their potential association with disc perforation.

MRI-based assessments will be performed using standardized imaging protocols, and all findings will be systematically recorded and evaluated. By integrating radiologic and clinical data, the study aims to improve the understanding of factors contributing to TMJ disc perforation and to support future diagnostic and therapeutic strategies.

ELIGIBILITY:
Inclusion Criteria:

* Patients with available temporomandibular joint (TMJ) MRI scans (both open- and closed-mouth)
* Age ≥14 years
* Complete clinical records including Visual Analogue Scale (VAS) pain scores and dental status
* Willingness to participate in the study and provide informed consent (for prospective studies)

Exclusion Criteria:

* Presence of systemic disorders affecting bone metabolism, including rheumatoid arthritis, chronic systemic corticosteroid therapy, Paget's disease, hypo- or hyperparathyroidism, osteomalacia, or renal osteodystrophy
* History of medications that could alter bone architecture
* Current orthodontic treatment
* History of head and neck trauma or surgery
* Presence of head and neck cystic or tumoral pathology
* Prior radiotherapy or chemotherapy
* Pregnancy
* Presence of ferromagnetic objects in the head (contraindication to MRI)

Ages: 14 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The study population will consist of approximately 282 patients (200 females and 82 males) aged 14-79 years who have undergone TMJ MRI scans for clinical evaluation. Patients will be included if they have complete MRI images (open- and closed-mouth) and corresponding clinical records, including Visual Analogue Scale (VAS) pain scores and detailed dental status. Individuals with systemic disorders affecting bone metabolism, history of bone-altering medications, current orthodontic treatment, prior head or neck trauma or surgery, head or neck cystic or tumoral pathology, previous radiotherapy or chemotherapy, pregnancy, or presence of ferromagnetic objects in the head will be excluded. The population will be stratified into two cohorts based on the presence or absence of TMJ disc perforation as determined by MRI.
Sampling Method: Probability Sample
Enrollment: 282 (Actual)
Dates: Start 2025-11-01 (Actual); Primary Completion 2025-12-03 (Actual); Study Completion 2025-12-03 (Actual)

PRIMARY OUTCOMES:
Presence of TMJ Disc Perforation | At MRI assessment (baseline, single time point)
  Dichotomous outcome (Yes/No) indicating the presence of temporomandibular joint disc perforation, determined from closed- and open-mouth MRI images assessed by an experienced radiologist/oral and maxillofacial surgeon.
  Unit of Measure: Percentage of joints with MRI-confirmed disc perforation

SECONDARY OUTCOMES:
Disc Configuration Distribution | At MRI assessment (baseline)
  Categorical outcome describing temporomandibular joint disc morphology classified as biconcave, concave, flattened, folded, amorphous, or perforated, determined from closed-mouth MRI images evaluated by an experienced radiologist/oral and maxillofacial surgeon.
  Unit of Measure: Percentage of joints in each disc morphology category
Disc Position (Closed/Open-mouth) | At MRI assessment (baseline)
  Categorical: Normal, Anterior Disc Displacement with Reduction (ADDWR), Anterior Disc Displacement without Reduction (ADDWoR). Determined by posterior band position relative to condyle on closed- and open-mouth images.
  Unit of Measure: Percentage of joints in each internal disc status category
Condylar Bone Marrow Signal Pattern | At MRI assessment (baseline)
  Categorical: Normal, Edema, Sclerosis, Combined Edema and Sclerosis. Proportion of joints with each signal pattern on PDWI and T2WI. Unit of Measure:
  Percentage of joints in each bone marrow signal pattern category
Joint Effusion Grade | At MRI assessment (baseline)
  Ordinal: Grade 0-3 on T2WI (Grade 0 = no effusion; Grade 1 = dot/linear; Grade 2 = bands; Grade 3 = accumulation). Distribution of effusion grades. Unit of Measure: Percentage of joints in each effusion grade
Pain Severity (VAS per TMJ) | At clinical assessment coincident with MRI (baseline): retrospective clinical data
  Continuous outcome describing temporomandibular joint pain intensity, measured using the Visual Analogue Scale (VAS; 0-10) as reported by patients and recorded by an oral and maxillofacial surgeon.
  Unit of Measure: Mean VAS pain score per joint (0-10)
Dental Status | At clinical assessment (baseline): retrospective clinical data
  Discrete outcome describing the number of missing permanent teeth, with individual tooth numbers recorded according to the dental charting system.
  Unit of Measure: Number of missing teeth per patient

CONTACTS AND LOCATIONS:
Locations (1):
- Recep Tayyip Erdoğan University Faculty of Dentistry, Rize, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No